CLINICAL TRIAL: NCT00286481
Title: A Double-Blind, Randomized, Placebo-Controlled Factorial Study to Evaluate the Efficacy and Safety of Lapaquistat and Simvastatin Alone and in Combination in Subjects With Hypercholesterolemia
Brief Title: Efficacy of Lapaquistat Acetate Alone or Combined With Simvastatin in Subjects With Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-475-020; U1111-1122-7978 (Registry Identifier: WHO)
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia; Drug Therapy
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lapaquistat Acetate 50 mg QD + Simvastatin (Experimental)
  Interventions: Drug: Lapaquistat acetate and simvastatin
- Lapaquistat Acetate 100 mg QD + Simvastatin (Experimental)
  Interventions: Drug: Lapaquistat acetate and simvastatin
- Simvastatin (Active Comparator)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Lapaquistat acetate and simvastatin — Lapaquistat acetate 50 mg, tablets, orally, once daily and stable dose of simvastatin for up to 12 weeks.
  Other Names: TAK-475; Zocor
  Arms: Lapaquistat Acetate 50 mg QD + Simvastatin
Drug: Lapaquistat acetate and simvastatin — Lapaquistat acetate 100 mg, tablets, orally, once daily and stable dose of simvastatin for up to 12 weeks.
  Other Names: TAK-475; Zocor
  Arms: Lapaquistat Acetate 100 mg QD + Simvastatin
Drug: Simvastatin — Lapaquistat acetate placebo-matching tablets, orally, once daily and stable dose of simvastatin for up to 12 weeks.
  Other Names: Zocor
  Arms: Simvastatin

SUMMARY:
The purpose of this study is to evaluate lapaquistat acetate, once daily (QD), taken alone or with simvastatin on cholesterol levels in treating patients with elevated cholesterol.

DETAILED DESCRIPTION:
Elevated plasma cholesterol (hypercholesterolemia) and various other plasma lipid imbalances (dyslipidemias) are major risk factors for coronary heart disease. Patients with hypercholesterolemia have elevated low-density lipoprotein cholesterol, which leads to atherosclerotic deposition of cholesterol in the arterial walls. As identified by the National Cholesterol Education Program Adult Treatment Panel III, lowering the low-density lipoprotein cholesterol plasma concentration effectively reduces cardiovascular morbidity and mortality and is essential for the prevention and management of coronary heart disease.

Currently, 3-hydroxy-3-methylglutaryl-coenzyme A reductase inhibitors (statins) are the first-line monotherapies prescribed to reduce low-density lipoprotein cholesterol, after diet and therapeutic lifestyle change. However, low doses of statins often fail to produce the ATP III-recommended levels of low-density lipoprotein cholesterol reduction, making it necessary to increase the dose or add an additional treatment. Dose increases of statins in turn may result in decreased tolerability and potential safety concerns which contribute to the high discontinuation rates of statins and their prescription at low, and often ineffective, doses.

The purpose of this study is to determine whether administration of lapaquistat acetate co-administered with simvastatin will be more efficacious in lowering low-density lipoprotein cholesterol, compared to lapaquistat or simvastatin alone. Total participation time in this study is anticipated to be 19 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Woman of childbearing potential can not to be pregnant, lactating, not planning on becoming pregnant, and agree to use acceptable forms of contraception throughout the course of the study.
* Prior to Randomization, has a low-density lipoprotein cholesterol level mean greater than or equal to 3.37 mmol/L and less than or equal to 5.70 mmol/L.
* Prior to Randomization, has a mean triglyceride level less than or equal to 4.52 mmol/L (400 mg/dL).
* Has clinical laboratory evaluations including clinical chemistry, hematology, and urinalysis within the defined reference range.

Exclusion Criteria:

* Has an alanine aminotransferase or aspartate aminotransferase level of greater than 1.5 times the upper limit of normal, active liver disease or jaundice.
* Has a serum creatinine of greater than 133 μmol/L.
* Has a creatine kinase greater than 3 times the upper limit of normal.
* Has type 1 or 2 diabetes mellitus.
* Has a previous history of cancer that had been in remission for less than 5 years prior to the first dose of study medication.
* Has an endocrine disorder, such as Cushing syndrome, hyperthyroidism, or inappropriately treated hypothyroidism, affecting lipid metabolism.
* Has a history of myocardial infarction, angina pectoris, transient ischemic attacks, cerebrovascular accident, peripheral vascular disease, abdominal aortic aneurysm, coronary revascularization or multiple factors that conferred a 10-year risk for coronary heart disease greater than 20% based on Framingham risk scoring.
* Has a positive hepatitis B surface antigen, or antibody to hepatitis C virus, as determined by medical history and/or subject's verbal report.
* Has a positive human immunodeficiency virus status or was taking antiretroviral medications, as determined by medical history.
* Has exposure to lapaquistat acetate in other studies, was participating in another investigational study, or had participated in an investigational study within the past 30 days or, for drugs with a long half-life, within a period of less than 5 times the drug's half-life. Has a known hypersensitivity or history of adverse reaction to simvastatin.
* Has a known hypersensitivity or history of adverse reaction to simvastatin.
* Has a history or presence of clinically significant food allergy that would prevent adherence to the recommended diet.
* Has a known heterozygous or homozygous familial hypercholesterolemia or known Type III hyperlipoproteinemia (familial dysbetalipoproteinemia).
* Has fibromyalgia, myopathy, rhabdomyolysis or unexplained muscle pain.
* Has uncontrolled hypertension
* Has inflammatory bowel disease, any other malabsorption syndrome, or had gastric bypass or any other surgical procedure for weight loss.
* Is unwilling or unable, in the opinion of the investigator, to comply with the protocol or scheduled appointments.
* Has a history of drug abuse or a history of alcohol abuse within the past 2 years.
* Has any other serious disease or condition that might reduced life expectancy, impaired successful management according to the protocol, or make the participant an unsuitable candidate to receive study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1362 (Actual)
Dates: Start 2006-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Low Density Lipoprotein cholesterol | Week 12 or Final Visit

SECONDARY OUTCOMES:
Adverse Events | Weeks: 2, 4, 8, and 12 or Final Visit
Physical Examination | Week 12 or Final Visit
Safety Laboratory Tests | Weeks: 2, 4, 8, and 12 or Final Visit
12- lead Electrocardiogram assessments | Week 12 or Final Visit
Best Corrected Visual Acuity results | Week 12 or Final Visit
Vital Signs | Weeks: 2, 4, 8, and 12 or Final Visit
Change from Baseline in Triglycerides | Week 12 or Final Visit
Change from Baseline in Total Cholesterol | Week 12 or Final Visit
Change from Baseline in High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in Very Low Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in apolipoprotein A1 | Week 12 or Final Visit
Change from Baseline in apolipoprotein B | Week 12 or Final Visit
Change from Baseline in non- High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in the ratio of Low Density Lipoprotein cholesterol/High Density | Week 12 or Final Visit
Change from Baseline in the ratio of Total Cholesterol/High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in the ratio of apolipoprotein A1/apolipoprotein B | Week 12 or Final Visit
Change from Baseline in high-sensitivity C-reactive protein | Week 12 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 2.59 mmol/L (100 mg/dL) | Week 12 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 3.37 mmol/L (130 mg/dL) | Week 12 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 4.14 mmol/L (160 mg/dL) | Week 12 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (67):
- United States (50):
  - Huntsville, Alabama
  - Chandler, Arizona
  - Scottsdale, Arizona
  - Sierra Vista, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - Long Beach, California
  - Sacramento, California
  - Spring Valley, California
  - Colorado Springs, Colorado
  - Hialeah, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Stuart, Florida
  - West Palm Beach, Florida
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Overland Park, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Edina, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Margate City, New Jersey
  - Raleigh, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Kettering, Ohio
  - Bartlesville, Oklahoma
  - Portland, Oregon
  - Beaver, Pennsylvania
  - Downingtown, Pennsylvania
  - Tipton, Pennsylvania
  - Goose Creek, South Carolina
  - Jackson, Tennessee
  - Nashville, Tennessee
  - San Antonio, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Lakewood, Washington
- Canada (17):
  - Abbotsford, British Columbia
  - Coquitlam, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Mount Pearl, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - Cornwall, Ontario
  - London, Ontario
  - Oakville, Ontario
  - Oshawa, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Cornwall, Prince Edward Island
  - Mirabel, Quebec
  - Saint-Lambert, Quebec
  - Sherbrooke, Quebec
  - Ste-Foy, Quebec

REFERENCES:
- [Result] Stein EA, Bays H, O'Brien D, Pedicano J, Piper E, Spezzi A. Lapaquistat acetate: development of a squalene synthase inhibitor for the treatment of hypercholesterolemia. Circulation. 2011 May 10;123(18):1974-85. doi: 10.1161/CIRCULATIONAHA.110.975284. Epub 2011 Apr 25. PMID 21518985